CLINICAL TRIAL: NCT02355145
Title: REALITY: A Non-inteRvEntional Study to Observe the rAtionaLe of selectIng add-on TherapY for Type 2 Diabetes Inadequately Controlled With Metformin in Real-life Practice at 1 Year Distance
Brief Title: Non-inteRvEntional Study to Observe rAtionaLe to Select add-on TherapY for Type 2 Diabetes Inadequately Controlled With Metformin.
Acronym: REALITY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00243
Record Dates: First submitted 2015-01-16; First posted 2015-02-04 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes, add-on diabetes therapy, rationale
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient group in moment 1 of evaluation: Study group enrolled in moment 1 of evaluation (Feb - Mar 2015)
- Patient group in moment 2 of evaluation: Study group enrolled in moment 2 of evaluation (Feb - Mar 2016) - 1 year distance from moment 1

SUMMARY:
A non-interventional, multicentre study to observe the main criteria used in clinical practice by physicians when selecting the second-line add-on therapy in patients with inadequately metformin-controlled type 2 diabetes in 2 time points at 1 year distance. Data will be collected by reviewing the medical records of patients with type 2 diabetes and add-on therapies at the time of presenting to endocrinologist according to clinical practice. The patients will participate in only one study visit, at the time of enrolment. Two study groups are to be defined at two time-points.

DETAILED DESCRIPTION:
A non-interventional, multicenter study to observe the main criteria used in clinical practice by physicians when selecting the second-line add-on therapy in patients with inadequately metformin-controlled type 2 diabetes in 2 time points at 1 year distance. The study will enrol a minimum of 500 patients in each time point, resulting in a total of at least 1000 from approximately 50 investigators from Bulgaria. Each investigator will recruit approximately 10 subjects.

The assignment of the patients to a particular add-on therapy is not decided in advance by the NIS protocol, but falls within current practice and the prescription of medicine is clearly separated from the decision to include the subject in the study. No additional diagnostic and monitoring procedures shall be applied to patients, other than daily clinical practice and the epidemiological methods shall be used for the analysis of collected data. The intention of the study is to collect data on patients with type 2 diabetes and add-on therapies under routine clinical care.

The patients will participate in only one study visit, at the time of enrolment, when they provide the written informed consent, thus allowing the access to their data. Data will be collected by reviewing the medical records of patients.

Two study groups are to be defined at each time-point - one study group enrolled in moment 1 of evaluation (Feb - Mar 2015) and one study group enrolled in moment 2 of evaluation (Feb - Mar 2016). A patient enrolled in study moment 1 may not be enrolled in study moment 2. No patient will be prospectively followed-up during the study.

Investigators participating in this non-interventional study will be diabetologists in outpatient settings, as this group of specialists treats most of the T2DM patients in Bulgaria.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent
* Female and/or male aged 18 years and over
* Diagnosis of type 2 diabetes mellitus
* Patients considered inadequately controlled with metformin with a current treatment based on any add-on diabetes therapy

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Current antidiabetes treatment with oral monotherapy
* Insulin treatment for type 2 diabetes
* Current participation in any clinical trial
* Patient who have been enrolled in the study at point 1 can not be enrolled at point 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients, inadequately controlled with metformin, with a current treatment based on any add-on (non-insulin) diabetes therapy.
Sampling Method: Probability Sample
Enrollment: 1005 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of usage by physicians of the main criteria for selecting the add-on therapy in patients with inadequately metformin-controlled type 2 diabetes | From moment 1 (up to 2 months from FSI) to moment 2 (1 year after moment 1)
  To describe and compare the main criteria used by physicians (regular outpatient setting) in selecting the add-on therapy in patients with inadequately metformin-controlled type 2 diabetes in 2 time points at 1 year distance. Descriptive analysis will be produced for the response to questions stratified by patients (binominal variable) and within physician clusters (derived percentages). To describe the overall changes descriptive analysis will be used for those physician who have responses both in 2 time points at 1 year distance.

SECONDARY OUTCOMES:
Number of years (duration) of add-on therapies in type 2 diabetes | in 2 time points at 1 year distance - moment 1 (up to 2 months from FSI) and moment 2 (1 year after moment 1)
  To describe the usage of add-on therapies in type 2 diabets and changes observed in 1 year. Descriptive analysis will be used within physician cluster for those physicians who have responses both in 2 time points at 1 year distance.
Percentage of subjects with specific comorbid conditions and/or diabetes complications | in 2 time points at 1 year distance - moment 1 (up to 2 months from FSI) and moment 2 (1 year after moment 1)
  To evaluate the prevalence of comorbidities and diabetes complications in study groups. Descriptive analysis will be produced within physician cluster.
Percentage of patients with target HbA1c level < 7% at the 2 time-points | in 2 time points at 1 year distance - moment 1 (up to 2 months from FSI) and moment 2 (1 year after moment 1)
  To evaluate the percentage if patients with target HbA1c level < 7% at the 2 time-points, by assessment of their last available HbA1c value. Descriptive analysis will be produced within physician cluster.
Number of years of type 2 diabetes disease duration | in 2 time points at 1 year distance - moment 1 (up to 2 months from FSI) and moment 2 (1 year after moment 1)
  To describe the characteristics of the disease at the time of initiating the add-on therapy in Bulgarian patients with type 2 diabetes. Descriptive analysis will be produced within physician cluster.
Frequency of the used classes of drugs | in 2 time points at 1 year distance - moment 1 (up to 2 months from FSI) and moment 2 (1 year after moment 1)
  To describe the usage of add-on therapies in type 2 diabets and changes observed in 1 year. Descriptive analysis will be used within physician cluster for those physicians who have responses both in 2 time points at 1 year distance.
Number of years until starting the add-on therapies after diagnosis | in 2 time points at 1 year distance - moment 1 (up to 2 months from FSI) and moment 2 (1 year after moment 1)
  To describe the characteristics of the disease at the time of initiating the add-on therapy in Bulgarian patients with type 2 diabetes. Descriptive analysis will be produced within physician cluster.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Staneva, Study Director — AstraZeneca Bulgaria
Locations (3):
- Bulgaria (3):
  - Research Site, Pleven
  - Research Site, Sofia
  - Research Site, Stara Zagora

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3768&filename=StudyReportSummaryD1843R00243.pdf